CLINICAL TRIAL: NCT04924478
Title: Evaluation of Volatile Organic Compound Signatures as a Predictive and Therapeutic Response Biomarker for Mepolizumab Therapy in Severe Eosinophilic Asthma
Brief Title: Evaluation of Volatile Organic Compounds in Mepolizumab Therapy
Acronym: EVOC4M
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: RHM MED1746
Record Dates: First submitted 2021-05-14; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Asthma; Eosinophilic
Keywords: Exhaled Breath; VOC; Mepolizumab; Severe Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum, blood, exhaled breath, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Asthma Patients Treated with Mepolizumab: Following treatment, patients will be stratified into responders or non-responders
  Interventions: Biological: Mepolizumab

INTERVENTIONS:
Biological: Mepolizumab — Patients will be receiving this treatment as part of their standard clinical care

SUMMARY:
This study will recruit patients who are being prescribed Mepolizumab as part of their standard clinical care for the treatment of severe eosinophilic asthma. Over the course of their treatment, research data (questionnaires) and research samples (blood, breath and urine) will be collected in parallel to standard clinical measurements.

The data and samples will be investigated to help better understand how Mepolizumab works, why it doesn't work in certain patients and why it works very well in others. This will help prescribers better identify patients that will benefit from Mepolizumab.

DETAILED DESCRIPTION:
EVOC4M is a prospective observational study investigating Mepolizumab in the treatment of severe eosinophilic asthma.

This study will recruit patients receiving Mepolizumab as part of their standard clinical care in an NHS commissioned Specialised Adult Severe Asthma Service. Over the course of their treatment, research data (questionnaires) and research samples (blood, breath and urine) will be collected in parallel to standard clinical measurements.

Clinical studies have demonstrated blood eosinophil levels to be predictive of the magnitude of the impact of Mepolizumab in reducing severe disease exacerbations but it is appreciated that there are still treatment failures despite this selection criteria. Clinical decision and policymaking are increasingly concerned by the health economic implications of these high-cost therapies and so clinical biomarkers are now being sought for theragnostics: prediction of treatment response

The study will try to identify biomarkers that will can discriminate between those that respond to Mepolizumab ("responders") and those that do not ("non-responders"). This will improve our understanding of how Mepolizumab works.

In particular, the investigators are interested in exhaled volatile organic compounds (VOCs), which are measured in exhaled breath samples. Exhaled breath is safe and easy to collect and has direct contact with the organ of interest, the airways. A VOC biomarker that predicts Mepolizumab success may translate to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years at Visit 1
* Able and willing to provide written informed consent and to comply with the study protocol
* Severe asthma confirmed after assessment by an asthma physician, requiring treatment with high dose inhaled corticosteroids (ICS) as per BTS criteria [≥1000 micrograms fluticasone propionate equivalent] and ≥ 1 additional drug for asthma [e.g. long acting beta2 agonist (LABA), leukotriene receptor antagonist (LTRA) such as montelukast, theophylline, long acting muscarinic antagonist (LAMA) such as tiotropium) at screening [participants may be included with a lower dose of current ICS at the discretion of the investigator if previous high ICS dose had led to side effects]
* Adherent with background asthma medication in the opinion of the local MDT
* Assessed and treatment optimized for any significant asthma-related co-morbidities in the opinion of the local MDT
* Considered suitable by an asthma specialist for treatment with a monoclonal antibody to block the Interleukin-5 pathway as per local practice, in accordance with NICE TA 431
* a recorded blood eosinophil count ≥0.3 x 109/L within the past year
* history of either ≥ 4 asthma exacerbations requiring high dose oral corticosteroids (exacerbations of asthma in the past year will be defined as worsening of asthma symptoms leading to treatment with prednisolone ≥30 mg oral corticosteroids for ≥3 days as defined by the ERS/ATS Task Force) OR
* has had continuous oral corticosteroids of at least the equivalent of prednisolone 5 mg per day over the previous 6 months

Exclusion Criteria:

* Acute exacerbation requiring high dose oral corticosteroids in the 4 weeks prior to Visit 1. Such patients would be re-assessed when 4 weeks clear of the oral corticosteroid course for re-screening.
* Long term systemic antibiotic or antifungal therapy
* Other clinically significant medical disease (including malignancy or immunodeficiency requiring treatment) or uncontrolled concomitant disease that is likely, in the opinion of the investigator, to require a change in therapy or impact the ability to participate in the study
* Active lung disease other than asthma [Note: Controlled obstructive sleep apnoea (OSA), minor bronchiectasis, asbestos pleural plaques or old (inactive) TB scars are not exclusion criteria]. Patients where an asthma-COPD overlap is suspected by the investigator are not eligible for inclusion
* History of current alcohol, drug, or chemical abuse or past abuse that would impair or risk the subject's full participation in the study, in the opinion of the investigator
* Current smoker or smoked in the past 12 month prior to Visit 1 or any history of e-cigarette use
* Female patients who are pregnant or lactating or planning a family
* Treatment with any of the following prior to Visit 1 or during the study
* Any biologic medicine for asthma or an immunomodulating biologic agent for other conditions in the 6 months prior to Visit 1
* An investigational agent within 30 days of Visit 1 (or five half-lives of the investigational agent, whichever is longer).
* Administration of live attenuated vaccine 30 days prior to Visit 1. Other types of vaccines are allowed.
* Other ongoing immunosuppressive/ immunomodulating therapy [e.g. methotrexate, ciclosporine, azathioprine] other than oral corticosteroids for asthma.
* Bronchial thermoplasty conducted within 6 months of Visit 1.
* Patients with helminth infections must be excluded until the infection has been treated
* Known hypersensitivity to Mepolizumab

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from University Hospital Southampton (UHS). UHS operates a regional specialist clinical severe asthma service, prescribing biological therapies, including Mepolizumab. Patients will be exclusively recruited from a pool of patients awaiting biological therapies for severe asthma at these centres. Patients are only eligible for Mepolizumab following NICE mandated multidisciplinary team approval reviewing biological eligibility, treatment adherence and satisfaction that other co-morbid conditions have been satisfactorily addressed.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Response to Mepolizumab | 12 months
  defined as positive if Clinical multidisciplinary team decision that patient has had a positive response OR >50% reduction in number of exacerbations per year OR 0.5 point reduction in ACQ score

OTHER OUTCOMES:
Change in Lung physiology with Mepolizumab therapy | 12 months
  measured by Impulse Oscillometry
Change in Immune responses with Mepolizumab therapy | 12 months
  measured by whole blood gene expression profiling

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Azim, MBBS, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Researchers and collaborators outside of the study team can submit a request to the PI to access study data at the end of the study for any ethical approved research or external collaborations.